CLINICAL TRIAL: NCT00814879
Title: A Pilot Randomized, Open-Label Study Comparing the Safety and Efficacy of a Raltegravir Based NRTI Sparing Regimen
Brief Title: Pilot Study of a Raltegravir Based NRTI Sparing Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Bristol-Myers Squibb (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0811004448; Yale-No Nukes
Record Dates: First submitted 2008-12-18; First posted 2008-12-25 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Acquired Immune Deficiency Syndrome; AIDS; Human Immunodeficiency Virus; HIV Infections
Keywords: Acquired Immune Deficiency Syndrome; AIDS; Anti-Infective Agents; Antiretroviral; Antiviral Agents; Atazanavir; Human Immunodeficiency Virus; HIV; HIV Protease Inhibitors; NRTI; Nucleoside Reverse Transcriptase Inhibitors; Raltegravir; Resistance; treatment experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Raltegravir Potassium; Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- a. (Active Comparator): N(t)RTI(s) based backbone & PI/r
  Interventions: Other: Standard treatment regimen
- b. (Experimental): Raltegravir (RAL) 400mg BID + atazanavir (ATV) 300 mg BID
  Interventions: Drug: Raltegravir; Drug: Atazanavir

INTERVENTIONS:
Drug: Raltegravir — 400 mg BID
  Other Names: Isentress
  Arms: b.
Drug: Atazanavir — 300 mg BID
  Other Names: Reyataz
  Arms: b.
Other: Standard treatment regimen — N(t)RTI(s) based backbone plus ritonavir boosted PI
  Arms: a.

SUMMARY:
This pilot study will provide data on the safety and efficacy of the combination of Raltegravir (RAL) 400mg BID + Atazanavir (ATV) 300 mg BID in Antiretroviral (ARV)-experienced subjects that have a suppressed HIV viral load on a Ritonavir (RTV) boosted Protease Inhibitor (PI) based regimen who are then switched to a regimen of RAL 400mg BID +ATV 300mg BID.

DETAILED DESCRIPTION:
The purpose of this pilot study is to compare the virological efficacy, as measured by the proportion of patients with plasma HIV-RNA below the limit of detection (<50 copies/mL), of two ARV regimens; patients are randomized to remain on regimens containing N(t)RTI(s) + PI/r or switch to Raltegravir + ATV but without N(t)RTI(s).

Study Arms:

1. N(t)RTI(s) based backbone + PI/r
2. Raltegravir (RAL) 400mg BID + atazanavir (ATV) 300 mg BID

Antiretroviral (ARV) treatment guidelines currently recommend ARV regimens containing a Nucleos(t)ide Reverse Transcriptase Inhibitors [N(t)RTI(s)] based backbone with a Non Nucleoside Reverse Transcriptase Inhibitor (NNRTI) or ritonavir boosted Protease Inhibitor (PI/r).(1) However, significant toxicity has been associated with N(t)RTI(s) and PI/r containing regimens. N(t)RTI(s) can cause lipoatrophy, lipid elevations, renal toxicity, neuropathy and lactic acidosis.(1) These toxicities have required clinicians and HIV-infected individuals to use alternative ARV regimens that do not use N(t)RTI(s). PIs are known to cause gastrointestinal side effects, dyslipidemia, and fat maldistribution (lipodystrophy).(1) The DHHS HIV treatment guidelines recommend that PIs should be given with a low dose of ritonavir (RTV). RTV is a PI that has an inhibitory effect on cytochrome P-450 3A4 isoenzyme which metabolizes most PIs. The addition of RTV serves as a pharmacokinetic "booster" by increasing PI drug concentrations.(1) However, RTV is known to increase PI side effects, elevate lipid levels and has significant drug-drug interactions with many medications given to HIV+ individuals.(1) These RTV drug interactions can complicate the medical care of an HIV-infected individual.

Raltegravir (RAL) is a recently FDA approved antiretroviral agent that inhibits HIV replication by blocking the integration of HIV proviral DNA into the host cell chromosomal DNA. RAL does not exhibit cross resistance to other ARV classes and thus has been initially used in HIV-infected individuals that are infected with drug resistant HIV strains. Recently published data on the use of RAL(2,3)in HIV-infected subjects with known ARV drug resistance or those without ARV drug resistance4 demonstrates that RAL is a potent agent, suppressing HIV viral loads in the majority of subjects and having excellent CD4 cell responses.(2-4) RAL is metabolized through glucuronidation by the uridine diphosphate-glucuronosyl transferase 1A1 (UGT1A1) enzyme pathway.(5)ATV is a known inhibitor of this enzyme pathway. ATV will increase RAL levels,(5) however, the current DHHS HIV treatment guidelines do not recommend a change in the dose of RAL if given with ATV as persons receiving ATV and RAL have demonstrated good tolerability of the combination and low side effect profiles.(1-3,5)

The availability of RAL provides an opportunity to examine alternative ARV strategies that may be equally efficacious and less toxic than those currently recommended in HIV treatment guidelines. Such combinations might include RAL+ATV regimen without a concomitant N(t)RTI(s) based backbone and/or the inclusion of RTV. However, there is little data available to date regarding such a combination. HIV care providers have already begun to use the combination of RAL+ unboosted ATV as the patients they care for are intolerant of RTV or have had major side effects/toxicity with N(t)NRTIs. More investigation is required to determine if RAL+ATV is an efficacious and safe alternative to RTV boosted PI based ARV strategies. Before a RAL based strategy that does not include N(t)RTIs or RTV can be compared to other ARV class strategies for long-term efficacy outcomes, preliminary data on a RAL+ATV based regimen is needed. This pilot study will provide data on the safety and efficacy of the combination of RAL 400mg BID + ATV 300 mg BID in ARV-experienced subjects that have a suppressed HIV viral load on a RTV boosted PI based regimen who are then switched to a regimen of RAL 400mg BID +ATV 300mg BID.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 positive
* On stable ARV-therapy for a minimum of 4 months with a HIV viral load of < 50 copies
* Currently on a N(t)RTI(s) based backbone + PI/r
* No prior history of PI drug resistance (by historical genotype or phenotype)
* Aged > 18 years of age
* Written informed consent
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

* Prior exposure to Raltegravir or Elvitegravir
* A detectable HIV viral load >50 copies within the last 4 months
* An ARV change within the last 4 months
* History of PI drug resistance
* Prior virologic failure on an ATV containing regimen
* Prior history of intolerance to ATV
* Pregnant or nursing mothers
* Pre-existing grade 3 or above laboratory toxicity except for lipids:
* Absolute neutrophil count (ANC) < 750 cells/mL.
* Hemoglobin < 8.0 g/dL.
* Platelet count < 50 000 cells/mL.
* AST, ALT and alkaline phosphatase > 5 x ULN.
* Serum bilirubin > 5 x ULN.
* calculated creatinine clearance of <50mL/min/1.73m2
* Patients with chronic active hepatitis B infection defined by positive serum Hbs antigen
* Use of any prohibited medications and/or the use of proton pump inhibitors in ATV plus RAL containing regimens)
* Patients with current alcohol or illicit substance use that in judgment of investigator makes study adherence unlikely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-05; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Kozal, MD, Principal Investigator — Yale University
Locations (5):
- United States (5):
  - Yale University School of Medicine, New Haven, Connecticut
  - Saint Raphael Healthcare System, New Haven, Connecticut
  - Waterbury Hospital, Waterbury, Connecticut
  - VA CT Healthcare Systems, West Haven, Connecticut
  - Comprehensive Care Center, Inc (dba Community AIDS Network), Sarasota, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 patients were randomized in this pilot study; 30 in each arm. Two patients randomized to stay on their N(t)NRTIs+PIr regimen were randomization failures as the patients did not for return for their baseline visit.
Groups:
- N(t)RTI(s) + PI/r: N(t)RTI(s) based backbone & PI/r
  Standard treatment regimen: N(t)RTI(s) based backbone plus ritonavir boosted PI
- RAL + ATV: Raltegravir (RAL) 400mg BID + atazanavir (ATV) 300 mg BID
  Raltegravir: 400 mg BID
  Atazanavir: 300 mg BID
Period: By Week 24
Arm/Group | N(t)RTI(s) + PI/r | RAL + ATV
Started | 28 | 30
Completed | 27 | 29
Not Completed | 1 | 1
Not completed — Cancer Diagnosis | 1 | 0
Not completed — Incarceration | 0 | 1
Period: By Week 48
Arm/Group | N(t)RTI(s) + PI/r | RAL + ATV
Started | 27 | 29
Completed | 25 | 26
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- N(t)NRTI + Plr: N(t)RTI(s) based backbone & PI/r
  Standard treatment regimen: N(t)RTI(s) based backbone plus ritonavir boosted PI
- Total: Total of all reporting groups
Arm/Group | N(t)NRTI + Plr | RAL + ATV | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (9.8) | 48.0 (9.7) | 48.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 23 | 24 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 21 | 20 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 30 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reaching Virologic Failure at Week 48.
Description: Virologic failure was defined by protocol as a plasma HIV RNA >50 c/mL on 2 consecutive occasions >7 days apart or > 10 000 c/mL on one occasion (in the absence of an intercurrent infection or recent immunization).
Time Frame: 48 Weeks
Measure: Number; unit: participants
Arm/Group | N(t)RTI(s) + PI/r | RAL + ATV
Number analyzed (Participants) | 25 | 26
participants | 2 | 3

2. Secondary Outcome: Number of Patients With < 400 Copies HIV RNA/mL at Week 48
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | N(t)RTI(s) + PI/r | RAL + ATV
Number analyzed (Participants) | 25 | 26
participants | 22 | 21

3. Secondary Outcome: CD4+ Cell Count
Time Frame: Weeks 24
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | N(t)NRTI + Plr | RAL + ATV
Number analyzed (Participants) | 27 | 29
cells/mm^3 | 599.4 (276.1) | 710.0 (37.80)

4. Secondary Outcome: CD4+ Cell Count
Time Frame: Week 48
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | N(t)RTI(s) + PI/r | RAL + ATV
Number analyzed (Participants) | 25 | 26
cells/mm^3 | 596.6 (289.1) | 665.9 (365.4)

5. Secondary Outcome: Cholesterol
Description: Total cholersterol (mg/dL)
Time Frame: baseline, week 24, week 48
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | N(t)RTI(s) + PI/r | RAL + ATV
Number analyzed (Participants) | 25 | 26
mg/dL
  Baseline | 166.25 (41.58) | 178.83 (46.97)
  Week 24 | 168.07 (43.77) | 169.65 (41.39)
  Week 48 | 167.41 (41.19) | 174.48 (37.12)

6. Secondary Outcome: Mean Change in Total Bilirubin (mg/dL) From Baseline
Description: mean change in total bilirubin from baseline
Time Frame: baseline and 48 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | N(t)RTI(s) + PI/r | RAL + ATV
Number analyzed (Participants) | 25 | 26
mg/dL | -0.15 (0.85) | 0.37 (1.39)

ADVERSE EVENTS:
Time Frame: Adverse events were assesses across the duration of the study through week 48.
Description: Serious adverse events were those that resulted in either hospitalization, death or pregnancy.
Arm/Group | N(t)RTI(s) + PI/r | RAL + ATV
Serious Adverse Events (participants affected / at risk) | 3/28 | 6/30
Other Adverse Events (participants affected / at risk) | 26/28 | 25/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N(t)RTI(s) + PI/r (N=28) | RAL + ATV (N=30)
Pregnancy (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (3)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric Panniculitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Death (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N(t)RTI(s) + PI/r (N=28) | RAL + ATV (N=30)
Anxiety (Psychiatric disorders) | 0 (0) | 4 (4)
CAP- Community Acquired Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 4 (6)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DOE- Dyspnea on Exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0)
Fever (Infections and infestations) | 1 (1) | 1 (1)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
GERD (Gastrointestinal disorders) | 2 (2) | 0 (0)
Headache (General disorders) | 1 (1) | 3 (3)
Myalgias (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Night Sweats (General disorders) | 1 (1) | 0 (0)
General Pain (General disorders) | 4 (7) | 3 (6)
Sinus Congestion (General disorders) | 1 (3) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 3 (4) | 3 (4)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Weight Loss (General disorders) | 1 (1) | 0 (0)
Other (General disorders) | 24 (77) | 24 (90) — Unspecified, non-serious, adverse events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes